CLINICAL TRIAL: NCT02122822
Title: Research for Immunotherapy of Glioblastoma With Autologous Heat Shock Protein gp96
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cure&Sure Biotech Co., LTD (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-TT-G-01
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Glioma
Keywords: supratentoria glioma
MeSH Terms: conditions — Glioma | interventions — glucose-regulated proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gp96 group (Experimental): autologous gp96 vaccination + basal treatment
  Interventions: Biological: gp96

INTERVENTIONS:
Biological: gp96 — vaccination of autologous gp96 derived from tumor tissue + basal treatment

SUMMARY:
RATIONALE: heat shock protein gp96-peptide complex made from a person's tumor cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This trial is studying the safety and effectiveness of autologous gp96 treatment of glioblastoma and to see how well it works in treating patients with newly diagnosed supratentoria glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the informed consent document; must sign the informed consent.
2. Aged 18 to 75 years old , sex is not limited
3. Newly Diagnosed supratentoria glioma, Must have undergone a at least a 80% resection
4. Availability of at least 1 g tumor sample.
5. Karnofsky functional status rating > or equal to 70.
6. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; Hemoglobin > 10g/dL ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase [AST], alanine amino transferase [ALT] <2.5 times institutional upper limit of normals [IULNs] ), and adequate renal function (BUN and creatinine <1.5 times IULNs)
7. Agree to Surgical indications of Heart & lung and without the coagulation system disease
8. Negative pregnancy test for female patients of childbearing potential
9. Agree to use contraception or abstain from sexual activity from the time of consent through 3 month after the end of study drug administration

Exclusion Criteria:

1. Inability to comply with study-related procedures
2. patient not suitable for Neurosurgery.
3. Unavailability of at least 6 doses of vaccine
4. Progression prior to vaccination as determined by the Principal Investigator
5. Patient with allergic constitution
6. Unstable or severe intercurrent medical conditions
7. Current diagnosis of Human Immunodeficiency Virus and Patients with active uncontrolled infection.
8. patients with any systemic disease needed to be treated with immunosuppressant or Corticosteroids.
9. any other clinical trials within 30 days pre-vaccination.
10. Female patients who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
blood count | baseline
  blood count within 3 days before first vaccination
blood count | within 3 days after the second injection
  blood count within 3 days after the second injection
blood count | within 3 days after the 6th injection
  blood count within 3 days after the 6th injection
blood chemistries | baseline
  blood chemistries test within 3 days before first vaccination
blood chemistries | within 3 days after the second injection
  blood chemistries test within 3 days after the second injection
blood chemistries | within 3 days after the 6th injection
  blood chemistries test within 3 days after the 6th injection
electrocardiogram | baseline
  electrocardiogram test within 3 days before first vaccination
electrocardiogram | within 3 days after the second injection
  electrocardiogram test within 3 days after the second injection
electrocardiogram | within 3 days after the 6th injection
  electrocardiogram test within 3 days after the 6th injection
progression-free survival rate of six month | six month after surgery
  progression-free survival rate of six month

SECONDARY OUTCOMES:
tumor control rate | six month after surgery
  tumor control rate at 6th month after surgery
progress free survive | up to 3 years
overall survive | up to 3 years
quality of life | up to 3 years
changes in antigen specific T cells | baseline and within 3 days before the 6th injection
  tumor antigen specific T cells was determined by IFN-γ Enzyme-linked immunosorbent spot using the autologous tumor cell lysis as the antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixian Gao, Doctor, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Affiliated to Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Ji N, Zhang Y, Liu Y, Xie J, Wang Y, Hao S, Gao Z. Heat shock protein peptide complex-96 vaccination for newly diagnosed glioblastoma: a phase I, single-arm trial. JCI Insight. 2018 May 17;3(10):e99145. doi: 10.1172/jci.insight.99145. eCollection 2018 May 17. PMID 29769450